CLINICAL TRIAL: NCT00969553
Title: A Phase I Single Dose Escalation Study of Two Dosing Schedules of BI 6727 Administered Intravenously in Asian Patients With Various Solid Cancers With Repeated Administration in Patients With Clinical Benefit
Brief Title: Dose Finding Study of BI 6727 (Volasertib) in Patients With Various Solid Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1230.16
Record Dates: First submitted 2009-08-31; First posted 2009-09-01 (Estimated); Results first posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-05

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — BI 6727

ARMS (1):
- BI 6727 (Experimental): Schedule A
  Interventions: Drug: BI 6727

INTERVENTIONS:
Drug: BI 6727 — Dose level 1

SUMMARY:
The primary objective of this trial is to identify the maximum tolerated dose (MTD) of BI 6727 in Asian cancer patients, and to provide safety data in terms of drug-related adverse events.

ELIGIBILITY:
Inclusion criteria:

1. Patients with histologically or cytologically confirmed diagnosis of advanced solid cancer
2. Age 18 years or older
3. Written informed consent
4. Eastern Cooperative Oncology Group (ECOG) performance score 2 or less

Exclusion criteria:

1. Serious illness or concomitant non-oncological disease.
2. Pregnancy or breast feeding
3. Active infectious disease
4. Absolute neutrophil count less than 1,500/cubic millimeter
5. Platelet count less than 100,000/cubic millimeter
6. Bilirubin greater than 1.5 mg/dL (> 26 µmol/L, SI unit equivalent)
7. Aspartate amino transferase (AST) and / or alanine amino transferase (ALT) greater than 2.5 times the upper limit of normal
8. Serum creatinine greater than 1.5x ULN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2009-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (2):
- Taiwan (2):
  - 1230.16.886002 Boehringer Ingelheim Investigational Site, Tainan
  - 1230.16.886001 Boehringer Ingelheim Investigational Site, Taipei

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A Phase I single dose escalation study of two dosing schedules of Volasertib administered intravenously in Asian patients with various solid cancers with repeated administration in patients with clinical benefit
Pre-assignment Details: Investigator notified the sponsor if a patient qualified for study participation. Sponsor informed the investigator about the respective treatment schedule and the dose tier. After completing dose level 1 of D1 schedule (i.e. 100mg), dose level 2 of D1 schedule (i.e. 200mg) and dose level 1 of D1+D8 schedule (50mg on Days 1+8,every 3 weeks) started
Groups:
- V 100 mg D1: A single dose of 100 milligram (mg) volasertib (V) on Day 1 every 3-week course. Volasertib was administered as a short infusion over 120 minutes (min) using an infusion pump.
  Immediately following the infusion of volasertib, the infusion tubing was washed with 100 millilitre (mL) physiological sodium chloride (0.9% NaCl) solution for a maximum duration of 10 min volasertib was administered strictly intravenous (i.v.).
- V 200 mg D1: A single dose of 200 mg volasertib on Day 1 every 3-week course. Volasertib was administered as a short infusion over 120 min using an infusion pump.
  Immediately following the infusion of volasertib, the infusion tubing was washed with 100 mL physiological sodium chloride (0.9% NaCl) solution for a maximum duration of 10 min volasertib was administered strictly i.v.
- V 250 mg D1: A single dose of 250 mg volasertib on Day 1 every 3-week course. Volasertib was administered as a short infusion over 120 min using an infusion pump.
  Immediately following the infusion of volasertib, the infusion tubing was washed with 100 mL physiological sodium chloride (0.9% NaCl) solution for a maximum duration of 10 min volasertib was administered strictly i.v.
- V 300 mg D1: A single dose of 300 mg volasertib on Day 1 every 3-week course. Volasertib was administered as a short infusion over 120 min using an infusion pump.
  Immediately following the infusion of volasertib, the infusion tubing was washed with 100 mL physiological sodium chloride (0.9% NaCl) solution for a maximum duration of 10 min volasertib was administered strictly i.v.
- V 350 mg D1: A single dose of 350 mg volasertib on Day 1 every 3-week course. Volasertib was administered as a short infusion over 120 min using an infusion pump.
  Immediately following the infusion of volasertib, the infusion tubing was washed with 100 mL physiological sodium chloride (0.9% NaCl) solution for a maximum duration of 10 min volasertib was administered strictly i.v.
- V 50 mg D1, D8: A single dose of 50 mg volasertib on Day 1 and Day 8 every 3-week course. Volasertib was administered as a short infusion over 120 min using an infusion pump. Immediately following the infusion of volasertib, the infusion tubing was washed with 100 mL physiological sodium chloride (0.9% NaCl) solution for a maximum duration of 10 min volasertib was administered strictly i.v.
- V 100 mg D1, D8: A single dose of 100 mg volasertib on Day 1 and Day 8 every 3-week course. Volasertib was administered as a short infusion over 120 min using an infusion pump. Immediately following the infusion of volasertib, the infusion tubing was washed with 100 mL physiological sodium chloride (0.9% NaCl) solution for a maximum duration of 10 min volasertib was administered strictly i.v.
- V 150 mg D1, D8: A single dose of 150 mg volasertib on Day 1 and Day 8 every 3-week course. Volasertib was administered as a short infusion over 120 min using an infusion pump. Immediately following the infusion of volasertib, the infusion tubing was washed with 100 mL physiological sodium chloride (0.9% NaCl) solution for a maximum duration of 10 min volasertib was administered strictly i.v.
- V 200 mg D1, D8: A single dose of 200 mg volasertib on Day 1 and Day 8 every 3-week course. Volasertib was administered as a short infusion over 120 min using an infusion pump. Immediately following the infusion of volasertib, the infusion tubing was washed with 100 mL physiological sodium chloride (0.9% NaCl) solution for a maximum duration of 10 min volasertib was administered strictly i.v.
Period: Overall Study
Arm/Group | V 100 mg D1 | V 200 mg D1 | V 250 mg D1 | V 300 mg D1 | V 350 mg D1 | V 50 mg D1, D8 | V 100 mg D1, D8 | V 150 mg D1, D8 | V 200 mg D1, D8
Started | 3 | 3 | 6 | 17 | 3 | 4 | 4 | 16 | 3
Completed | 0 | 0 | 0 | 1 (on-treatment at analysis data base lock date (27-Oct-2011)) | 0 | 0 | 0 | 2 (on-treatment at analysis data base lock date (27-Oct-2011)) | 0
Not Completed | 3 | 3 | 6 | 16 | 3 | 4 | 4 | 14 | 3
Not completed — Progressive disease (PD) | 2 | 2 | 6 | 9 | 2 | 4 | 2 | 12 | 3
Not completed — Dose limiting Toxicity (DLT) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Refused cont. medication | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Not completed — Not specified above | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The treated set consisted of all patients who received at least one dose of volasertib.
Groups:
- V100 D1: A single dose of 100 mg volasertib on Day 1 every 3-week course.
- V200 D1: A single dose of 200 mg volasertib on Day 1 every 3-week course.
- V250 D1: A single dose of 250 mg volasertib on Day 1 every 3-week course.
- V300 D1: A single dose of 300 mg volasertib on Day 1 every 3-week course.
- V350 D1: A single dose of 350 mg volasertib on Day 1 every 3-week course.
- V50 D1, D8: A single dose of 50 mg volasertib on Day 1 and Day 8 every 3-week course.
- V100 D1, D8: A single dose of 100 mg volasertib on Day 1 and Day 8 every 3-week course.
- V150 D1, D8: A single dose of 150 mg volasertib on Day 1 and Day 8 every 3-week course.
- V200 D1, D8: A single dose of 200 mg volasertib on Day 1 and Day 8 every 3-week course.
- Total: Total of all reporting groups
Arm/Group | V100 D1 | V200 D1 | V250 D1 | V300 D1 | V350 D1 | V50 D1, D8 | V100 D1, D8 | V150 D1, D8 | V200 D1, D8 | Total
Number analyzed (Participants) | 3 | 3 | 6 | 17 | 3 | 4 | 4 | 16 | 3 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (8.0) | 55.7 (9.3) | 52.0 (4.7) | 53.4 (11.4) | 52.3 (9.1) | 48.5 (8.5) | 51.5 (18.2) | 60.2 (10.0) | 66.7 (3.1) | 56.2 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 3 | 5 | 2 | 2 | 2 | 7 | 1 | 24
  Male | 2 | 2 | 3 | 12 | 1 | 2 | 2 | 9 | 2 | 35

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Dose Limiting Toxicities (DLT) in Cycle 1 for the Determination of the Maximum Tolerated Dose (MTD) of Volasertib
Description: Primary objective for this trial was to identify the MTD of volasertib for 2 dosing schedules. The MTD was defined as the highest volasertib dose studied for which the incidence of DLT was less than 2/6 patients. The MTD was defined on the basis of DLTs observed during the first treatment course only. In this outcome measure the percentage of participants with DLTs in cycle 1 is presented.
Time Frame: From first administration of study drug up to 3 weeks
Population: The treated set consisted of all patients whe received at least one dose of volasertib.
Measure: Number; unit: percentage of participants
Arm/Group | V100 D1 | V200 D1 | V250 D1 | V300 D1 | V350 D1 | V50 D1, D8 | V100 D1, D8 | V150 D1, D8 | V200 D1, D8
Number analyzed (Participants) | 3 | 3 | 6 | 17 | 3 | 4 | 4 | 16 | 3
percentage of participants | 0.0 | 0.0 | 16.7 | 23.5 | 100 | 0.0 | 0.0 | 0.0 | 66.7

2. Primary Outcome: MTD of Volasertib
Description: Primary objective for this trial was to identify the MTD of volasertib for 2 dosing schedules. The MTD was defined as the highest volasertib dose studied for which the incidence of DLT was less than 2/6 patients. This outcome measure shows the MTD.
Time Frame: From the first administration of study drug up to 3 weeks
Population: The treated set.
Measure: Number; unit: milligram (mg)
Groups:
- Volasertib D1 Schedule: A single dose of volasertib on Day 1 every 3-week course.
- Volasertib D1 and D 8 Schedule: A single dose of volasertib on Day 1 and Day 8 every 3-week course.
Arm/Group | Volasertib D1 Schedule | Volasertib D1 and D 8 Schedule
Number analyzed (Participants) | 17 | 16
milligram (mg) | 300 | 150

3. Secondary Outcome: Percentage of Participants With Incidence and Intensity of Drug-related AEs According to CTCAE v.3.0
Description: Percentage of participants with incidence and intensity of drug-related AEs according to Common Terminology Criteria for Adverse Events (CTCAE) v.3.0. This endpoint will be presented as a percentage of patients with adverse event by treatment and the highest CTCAE grade of the related AE.
Time Frame: From first administration of volasertib to 21 days after the last dose, up to 548 days
Population: Treated Set
Measure: Number; unit: Percentage of participants
Arm/Group | V100 D1 | V200 D1 | V250 D1 | V300 D1 | V350 D1 | V50 D1, D8 | V100 D1, D8 | V150 D1, D8 | V200 D1, D8
Number analyzed (Participants) | 3 | 3 | 6 | 17 | 3 | 4 | 4 | 16 | 3
Percentage of participants
  CTCAE Grade 1 | 0.0 | 0.0 | 0.0 | 5.9 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  CTCAE Grade 2 | 0.0 | 66.7 | 33.3 | 11.8 | 0.0 | 25.0 | 50.0 | 43.8 | 0.0
  CTCAE Grade 3 | 33.3 | 0.0 | 16.7 | 35.3 | 0.0 | 0.0 | 0.0 | 18.8 | 33.3
  CTCAE Grade 4 | 0.0 | 0.0 | 33.3 | 29.4 | 100.0 | 0.0 | 0.0 | 6.3 | 66.7
  CTCAE Grade 5 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

4. Secondary Outcome: Change From Baseline to Last Value on Treatment in Platelets
Description: This endpoint will be presented as a change from baseline to last value on treatment in platelets.
Time Frame: Baseline (Visit 1, prior to first administration of volasertib) and up to 21 days after last observation on treatment (up to 548 days)
Population: Treated Set
Measure: Mean (Standard Deviation); unit: 10^9 platelets/ Litre (L)
Arm/Group | V100 D1 | V200 D1 | V250 D1 | V300 D1 | V350 D1 | V50 D1, D8 | V100 D1, D8 | V150 D1, D8 | V200 D1, D8
Number analyzed (Participants) | 3 | 3 | 6 | 17 | 3 | 4 | 4 | 16 | 3
10^9 platelets/ Litre (L) | -30 (48) | -62 (30) | -5 (114) | -10 (173) | -55 (150) | -18 (29) | -69 (29) | -94 (111) | 42 (119)

5. Secondary Outcome: Change From Baseline to Last Value on Treatment in Neutrophils
Description: This endpoint will be presented as a change from baseline to last value on treatment in neutrophils.
Time Frame: as for outcome 4
Population: Treated Set
Measure: Mean (Standard Deviation); unit: 10^9 neutrophils / Litre (L)
Arm/Group | V100 D1 | V200 D1 | V250 D1 | V300 D1 | V350 D1 | V50 D1, D8 | V100 D1, D8 | V150 D1, D8 | V200 D1, D8
Number analyzed (Participants) | 3 | 3 | 6 | 17 | 3 | 4 | 4 | 16 | 3
10^9 neutrophils / Litre (L) | 0.9 (3.4) | -1.4 (1.1) | -1.3 (1.9) | -0.8 (3.2) | -0.7 (3.2) | 1.3 (1.4) | 1.0 (4.4) | -1.4 (2.6) | 3.1 (6.4)

6. Secondary Outcome: Patient Performance
Description: This endpoint will present the best clinical assessment. The investigator will perform a clinical assessment. An evaluation will be done whether the patient appears to be clinically improved, unchanged, or deteriorated. The presented numbers show the percentage of patients.
Time Frame: From first administration of volasertib to the last dose, up to 527 days
Population: Treated Set
Measure: Number; unit: percentage of participants
Arm/Group | V100 D1 | V200 D1 | V250 D1 | V300 D1 | V350 D1 | V50 D1, D8 | V100 D1, D8 | V150 D1, D8 | V200 D1, D8
Number analyzed (Participants) | 3 | 3 | 6 | 17 | 3 | 4 | 4 | 16 | 3
percentage of participants
  Unknown | 0 (48) | 0 (30) | 0 (114) | 6 (173) | 0 (150) | 0 (29) | 0 (29) | 0 (111) | 0 (119)
  Improved | 0 | 0 | 0 | 6 | 67 | 25 | 0 | 13 | 0
  Unchanged | 100 | 100 | 100 | 88 | 33 | 50 | 75 | 81 | 100
  Deteriorated | 0 | 0 | 0 | 0 | 0 | 25 | 25 | 6 | 0

7. Secondary Outcome: Vital Signs (Blood Pressure)
Description: This endpoint will be presented as a change from baseline at last observation of systolic blood pressure (SBP), diastolic blood pressure (DBP) in millimeter of mercury (mmHg) and pulse rate (PR) in beats per minute (bpm). In this outcome measure SBP and DBP are presented.
Time Frame: Baseline (Visit 1, prior to the first administration of volasertib), up to 21 days after last observation on treatment (up to 548 days)
Population: Treated Set
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | V100 D1 | V200 D1 | V250 D1 | V300 D1 | V350 D1 | V50 D1, D8 | V100 D1, D8 | V150 D1, D8 | V200 D1, D8
Number analyzed (Participants) | 3 | 3 | 6 | 17 | 3 | 4 | 4 | 16 | 3
mmHg
  SBP, chg from baseline at last observation | -19.0 (19.5) | 4.7 (14.2) | 0.0 (8.3) | -1.0 (19.1) | -12.3 (10.8) | 6.0 (12.7) | 1.5 (11.0) | -8.9 (16.9) | -3.3 (7.6)
  DBP, chg from baseline at last observation | -4.0 (9.0) | 2.0 (5.0) | -1.3 (11.3) | -1.9 (11.3) | -7.7 (10.0) | 10.3 (9.0) | 2.3 (10.4) | -2.9 (8.2) | 1.0 (6.2)

8. Secondary Outcome: Vital Signs (Pulse Rate)
Description: This endpoint will be presented as a change from baseline at last observation of systolic blood pressure (SBP), diastolic blood pressure (DBP) in millimeter of mercury (mmHg) and pulse rate (PR) in beats per minute (bpm). In this outcome measure the pulse rate is presented.
Time Frame: as for outcome 7
Population: Treated Set
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | V100 D1 | V200 D1 | V250 D1 | V300 D1 | V350 D1 | V50 D1, D8 | V100 D1, D8 | V150 D1, D8 | V200 D1, D8
Number analyzed (Participants) | 3 | 3 | 6 | 17 | 3 | 4 | 4 | 16 | 3
bpm | 18.3 (10.3) | 9.7 (15.5) | 16.5 (5.8) | 10.4 (16.5) | 2.7 (12.1) | 13.5 (7.0) | 10.0 (5.0) | 5.1 (18.9) | 12.7 (8.5)

9. Secondary Outcome: ECG
Description: This endpoint will be presented as a change from individual baseline in QT interval, corrected according to Fridericias formula (QTcF) to end of infusion (2 hours) and 24 hours after first infusion in Cycle 1.
Time Frame: Baseline, 2 hours (before the end of infusion of volasertib) and 24 hours after first infusion in Cycle 1
Population: Treated Set, only the patients in the Maximum Tolerated Dose (MTD) groups are evaluated for this endpoint.
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Arm/Group | V300 D1 | V150 D1, D8
Number analyzed (Participants) | 17 | 16
milliseconds (ms)
  Change from baseline after 2 hours | 21.0 (10.6) | 13.9 (7.7)
  Change from baseline after 24 hours | 5.2 (10.4) | 6.3 (9.7)

10. Secondary Outcome: Objective Response
Description: The objective response (OR) was defined as complete response (CR; disappearance of all target lesions) or partial response (PR; at least a 30 percent decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest) assessed by tumour measurement and evaluated according to the Response Evaluation Criteria in solid tumours (RECIST), version 1.0.
  The data represents the percentage of patients.
Time Frame: At screening and at the end of every other treatment course up to 527 days (= longest treatment exposure)
Population: The treated set
Measure: Number; unit: percentage of patients
Arm/Group | V100 D1 | V200 D1 | V250 D1 | V300 D1 | V350 D1 | V50 D1, D8 | V100 D1, D8 | V150 D1, D8 | V200 D1, D8
Number analyzed (Participants) | 3 | 3 | 6 | 17 | 3 | 4 | 4 | 16 | 3
percentage of patients
  OR: no or unknown | 100 | 100 | 100 | 100 | 67 | 100 | 100 | 94 | 100
  OR: yes | 0 | 0 | 0 | 0 | 33 | 0 | 0 | 6 | 0

11. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) is defined as the duration of time from start of treatment to time of progression or death. PFS was assessed by tumour measurement and evaluated according to RECIST, version 1.0.
Time Frame: At screening and at the end of every other treatment course up to 527 days (= longest treatment exposure)
Population: The treated set
Measure: Median (Full Range); unit: days
Arm/Group | V100 D1 | V200 D1 | V250 D1 | V300 D1 | V350 D1 | V50 D1, D8 | V100 D1, D8 | V150 D1, D8 | V200 D1, D8
Number analyzed (Participants) | 3 | 3 | 6 | 17 | 3 | 4 | 4 | 16 | 3
days | 83.0 [48 to 211] | 62.0 [37 to 84] | 48.0 [43 to 82] | 49.0 [30 to 139] | 274.0 [49 to 274] | 42.5 [8 to 254] | 92.0 [8 to 267] | 58.0 [8 to 499] | 45.0 [43 to 56]

12. Secondary Outcome: Response Duration
Description: The duration of overall response was measured from the time measurement criteria were met for complete response (CR) or partial response (PR), whichever was recorded first, until the first date that recurrent or progressive disease was objectively documented. The duration of overall CR was measured from the time measurement criteria were first met for CR until the first date that recurrent disease was objectively documented.
Time Frame: From first drug administration up to at 3 month interval after final End of treatment visit until disease progression, death, or lost to follow-up, up to 548 days
Population: The reason not to analyze the duration of objective response is that only 2 patients in different arms achieved an objective response and the analysis would reduce to a single patient case report.
Arm/Group | V100 D1 | V200 D1 | V250 D1 | V300 D1 | V350 D1 | V50 D1, D8 | V100 D1, D8 | V150 D1, D8 | V200 D1, D8
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Disease Control
Description: The disease control (DC) presented are the percentage of patients with CR, PR or stable disease as best response throughout the study assessed by tumour measurement and evaluated according to RECIST, version 1.0.
Time Frame: At screening and at the end of every other treatment course up to 527 days (= longest treatment exposure)
Population: The treated set
Measure: Number; unit: percentage of patients
Arm/Group | V100 D1 | V200 D1 | V250 D1 | V300 D1 | V350 D1 | V50 D1, D8 | V100 D1, D8 | V150 D1, D8 | V200 D1, D8
Number analyzed (Participants) | 3 | 3 | 6 | 17 | 3 | 4 | 4 | 16 | 3
percentage of patients
  DC: no or unknown | 33 | 33 | 67 | 59 | 33 | 75 | 50 | 38 | 100
  DC: yes | 67 | 67 | 33 | 41 | 67 | 25 | 50 | 63 | 0

14. Secondary Outcome: Sum of the Largest Diameters of Target Lesions
Description: The individual time profile of the sum of the largest diameters of target lesions (LD) is presented graphically for each patient in the Clinical Trial Report (CTR) only. No descriptive statistics were planned.
Time Frame: At screening and at the end of every other treatment course up to 527 days (= longest treatment exposure)
Population: No descriptive statistics were calculated, but the time profile of sum of largest diameter was plotted for each patient.
Arm/Group | V100 D1 | V200 D1 | V250 D1 | V300 D1 | V350 D1 | V50 D1, D8 | V100 D1, D8 | V150 D1, D8 | V200 D1, D8
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Pharmacokinetics (PK) AUC0-∞ of Volasertib
Description: The PK of volasertib will be presented for the area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) for the population attending the D1 schedule, the area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to 168 hours (AUC0-168) for the population attending the D1+ D8 schedule and the maximum measured concentration of volasertib in plasma (Cmax). In this outcome measure AUC0-∞ is presented.
Time Frame: Both schedules: 10 minutes prior to first drug administration and 1 hour (h), 2, 2:30, 3, 4, 8, 24, 336h thereafter; additional planned times in schedule D1+D8: 167:50, 169, 170, 170:30, 171, 172, 176, 192h; additional planned time in D1 schedule: 168h
Population: Treated Set. All evaluable patients were included in the PK analyses. Patients who were considered not evaluable were not included. A patient was considered to be not evaluable if they had an important protocol violation relevant to the evaluation of PK, or they had insufficient data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: in nanogram*hours/millilitre (ng*h/mL)
Arm/Group | V100 D1 | V200 D1 | V250 D1 | V300 D1 | V350 D1
Number analyzed (Participants) | 3 | 3 | 5 | 16 | 2
in nanogram*hours/millilitre (ng*h/mL) | 2140 (15.9) | 3280 (28.6) | 6140 (38.9) | 6260 (40.3) | 9790 (14.6)

16. Secondary Outcome: Pharmacokinetics (PK) AUC0-168 of Volasertib
Description: The PK of volasertib will be presented for the area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) for the population attending the D1 schedule, the area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to 168 hours (AUC0-168) for the population attending the D1+ D8 schedule and the maximum measured concentration of volasertib in plasma (Cmax). In this outcome measure AUC0-168 is presented.
Time Frame: as for outcome 15
Population: Treated Set. All evaluable patients were included in the PK analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: in nanogram*hours/millilitre (ng*h/mL)
Arm/Group | V50 D1, D8 | V100 D1, D8 | V150 D1, D8 | V200 D1, D8
Number analyzed (Participants) | 3 | 2 | 14 | 2
in nanogram*hours/millilitre (ng*h/mL)
  AUC0-168, 1st infusion | 590 (20.8) | 1380 (1.01) | 1890 (54.4) | 3320 (0.317)
  AUC0-168, 2nd infusion | 847 (16.7) | 1870 (19.8) | 2620 (67.1) | 4300 (16.0)

17. Secondary Outcome: Pharmacokinetics (PK) Cmax of Volasertib
Description: The PK of volasertib will be presented for the area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) for the population attending the D1 schedule, the area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to 168 hours (AUC0-168) for the population attending the D1+ D8 schedule and the maximum measured concentration of volasertib in plasma (Cmax). In this outcome measure Cmax is presented.
Time Frame: as for outcome 15
Population: Treated Set. All evaluable patients were included in the PK analyses. Patients who were considered not evaluable were not included. A patient was considered to be not evaluable if they had an important protocol violation relevant to the evaluation of PK, or they had insufficient data. D1 Schedule, no administration of trial drug on Day 8.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | V100 D1 | V200 D1 | V250 D1 | V300 D1 | V350 D1 | V50 D1, D8 | V100 D1, D8 | V150 D1, D8 | V200 D1, D8
Number analyzed (Participants) | 3 | 3 | 5 | 16 | 3 | 4 | 3 | 15 | 3
ng/mL
  After infusion Day 1 | 186 (7.87) | 540 (31.5) | 540 (37.0) | 489 (33.1) | 675 (3.19) | 106 (67.3) | 234 (2.99) | 235 (32.5) | 410 (22.1)
  After infusion Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 14 | 2
  After infusion Day 8 |  |  |  |  |  | 104 (47.6) | 212 (31.9) | 240 (49.4) | 431 (1.15)

ADVERSE EVENTS:
Time Frame: From inclusion into the study to 21 days after last drug administration (up to 548 days)
Arm/Group | V100 D1 | V200 D1 | V250 D1 | V300 D1 | V350 D1 | V50 D1, D8 | V100 D1, D8 | V150 D1, D8 | V200 D1, D8
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 2/6 | 7/17 | 1/3 | 0/4 | 2/4 | 7/16 | 2/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 17/17 | 3/3 | 3/4 | 4/4 | 16/16 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | V100 D1 (N=3) | V200 D1 (N=3) | V250 D1 (N=6) | V300 D1 (N=17) | V350 D1 (N=3) | V50 D1, D8 (N=4) | V100 D1, D8 (N=4) | V150 D1, D8 (N=16) | V200 D1, D8 (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Device occlusion (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Liver abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | V100 D1 (N=3) | V200 D1 (N=3) | V250 D1 (N=6) | V300 D1 (N=17) | V350 D1 (N=3) | V50 D1, D8 (N=4) | V100 D1, D8 (N=4) | V150 D1, D8 (N=16) | V200 D1, D8 (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 5 | 7 | 3 | 1 | 1 | 6 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 3 | 13 | 2 | 0 | 2 | 6 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 12 | 3 | 1 | 1 | 6 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 3 | 12 | 3 | 0 | 1 | 1 | 2
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 4 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 2 | 1 | 0 | 1 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 5 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroduodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 4 | 2 | 0 | 1 | 4 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Reflux oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 2 | 3 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 2
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0
Device occlusion (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 3 | 5 | 1 | 0 | 1 | 1 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 1 | 1 | 2 | 1 | 0 | 1 | 1 | 1
Pain (General disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 2 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 4 | 1 | 1 | 1 | 2 | 1
Tenderness (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Penis injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Electrocardiogram QRS complex abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 2 | 4 | 0 | 1 | 0 | 3 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 3 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 2 | 1 | 1 | 2 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Scrotal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 3 | 1 | 1 | 1 | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 3 | 3 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 3 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.